CLINICAL TRIAL: NCT01178671
Title: Combined Mirtazapine and Selective Serotonin Reuptake Inhibitor (SSRI) Treatment of Post-traumatic Stress Disorder (PTSD)
Brief Title: Combined Mirtazapine and SSRI Treatment of PTSD: A Placebo-Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Franklin Schneier, Research Psychiatrist, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34MH091336 (NIH); R34MH091336 (NIH)
Record Dates: First submitted 2010-07-29; First posted 2010-08-10 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; trauma; anxiety disorder; medication; sertraline; mirtazapine; pharmacotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Anxiety Disorders | interventions — Mirtazapine; Sertraline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertraline and Mirtazapine (Experimental): Flexible dose of both medications for up to 24 weeks
  Interventions: Drug: Mirtazapine; Drug: Sertraline
- Sertraline and Sugar pill (Active Comparator): Sertraline and Sugar pill for up to 24 weeks
  Interventions: Drug: Sertraline; Other: Sugar pill

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine capsule, flexible dose of 15-45 mg/day for up to 24 weeks
  Other Names: Remeron
  Arms: Sertraline and Mirtazapine
Drug: Sertraline — Sertraline tablet, flexible dose of 25-200mg/day for up to 24 weeks
  Other Names: Zoloft
Other: Sugar pill — Sugar pill capsule, flexible dose of 1-3 per day, for up to 24 weeks
  Other Names: placebo
  Arms: Sertraline and Sugar pill

SUMMARY:
The overall goal of this study is to examine the efficacy of the combination of mirtazapine and sertraline in the treatment of posttraumatic stress disorder (PTSD). Sertraline is FDA-approved for PTSD, but it is often not fully effective. The combination of mirtazapine and serotonin reuptake inhibitors like sertraline has appeared highly effective in a related disorder -- depression.

In this study, sixty patients with chronic PTSD will be randomized to treatment with either sertraline + mirtazapine or sertraline + placebo for 12 weeks. Patients who show at least a minimal response after 12 weeks will continue for another 12 weeks on the same treatment.

DETAILED DESCRIPTION:
This double-blind randomized controlled trial was conducted from January 2011 to February 2014. To acquire a diverse sample, outpatients were recruited at an academic medical center and at a private mental health clinic with primarily Spanish-speaking patients. A single team of investigators conducted the trial at both settings. Individuals with chronic PTSD were randomly assigned to 24 weeks of double-blind treatment with sertraline plus mirtazapine or sertraline plus placebo. This study was conducted in compliance with the Code of Ethics of the World Medical Association (Declaration of Helsinki) and the standards established by an Institutional Review Board and by the National Institutes of Health. Informed consent was obtained from participants after the nature of the procedures was explained.

Participants Participants were adults ages 18-75, referred by clinicians or responding to advertisements. After a preliminary telephone screening, eligibility was determined by clinical interview and confirmed by structured interview with trained raters using the Clinician-Administered PTSD Scale (CAPS) and the Structured Clinical Interview for DSM-IV Axis I Disorders -- Patient Edition. Participants had a principal Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnosis of chronic PTSD of at least moderate severity (CAPS score ≥50), and English or Spanish fluency. Bilingual clinicians treated and assessed individuals with Spanish language preference. Exclusion criteria were significant suicidal ideation; lifetime psychotic disorder, bipolar disorder, organic mental disorder, or seizure disorder; alcohol or substance use disorder in the past 3 months; unstable medical illness; history of traumatic brain injury of greater than moderate severity; pregnancy or nursing; unwillingness to use contraception (for women of childbearing potential); prior nonresponse to sertraline or combined treatment, or intolerance of sertraline or mirtazapine); and psychotropic medication use during the prior 2 weeks (4 weeks for monoamine oxidase inhibitors or fluoxetine), except that zolpidem for insomnia was allowed up to three times per week during the week prior to randomization; psychotherapy initiated within 3 months before randomization. Concomitant psychotropic medications were not permitted during the study.

Randomization and Blinding Randomization used randomly permuted blocks stratified by patient language preference (English vs. Spanish), implemented by the data manager who had no patient contact. Mirtazapine 15 mg capsules or matching placebo capsules were packaged by a pharmacist with no patient contact. Patients were reminded at each visit with the independent evaluator (IE) to not discuss medication or adverse events, and allocations were concealed from all research personnel throughout each patient's participation.

Treatments A single psychiatrist saw each patient for medication management, with an initial visit of 45 minutes and subsequent 30 minute visits weekly for two weeks, biweekly through week 12, then at 4-week intervals. At each visit the psychiatrist assessed clinical improvement and adverse events. Mirtazapine/placebo was initiated at 30 mg (two capsules) at bedtime for four weeks, after which patients without significant adverse events and with persistent PTSD symptoms had dose increased to a maximum of 45 mg/day. Dose could be decreased for intolerable adverse events, to a minimum of 15mg/day. Sertraline was initiated at 25 mg/day for four days, then increased as tolerated to 50 mg/day for the remainder of Week 1, 100 mg/day for Weeks 2-4, 150 mg/d for Weeks 5-6, and then 200 mg/day. Dosage could be decreased as clinically indicated to a minimum of 50 mg/day. Compliance was assessed with patient diaries and pill counts.

Patients who prematurely discontinued study medication were encouraged to return for all assessments through week 24.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of chronic PTSD
* Fluent in English or Spanish

Exclusion Criteria:

* Past or current schizophrenia, schizoaffective disorder, organic mental disorder, bipolar disorder, or antisocial personality disorder.
* Substance abuse of dependence diagnosis in past 3 months
* Suicidal ideation or behavior in past 6 months that poses a significant danger.
* Medical illness that could significant increase risk of sertraline and mirtazapine treatment or assessment of response
* History of traumatic brain injury of greater than mild severity
* History of seizure disorder (except febrile seizure in childhood)
* Currently taking medication which has been effective for patient's PTSD.
* Inability to tolerate or unwillingness to accept a drug-free period prior to beginning the study for certain psychiatric medications.
* History of inability to tolerate sertraline or mirtazapine or inadequate response to an adequate trial of combined treatment.
* Pregnancy, lactation; for women of childbearing potential, not using an effective birth control method.
* Current cognitive-behavioral therapy. Any psychotherapy initiated within 3 months of beginning this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Anxiety Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneier FR, Campeas R, Carcamo J, Glass A, Lewis-Fernandez R, Neria Y, Sanchez-Lacay A, Vermes D, Wall MM. COMBINED MIRTAZAPINE AND SSRI TREATMENT OF PTSD: A PLACEBO-CONTROLLED TRIAL. Depress Anxiety. 2015 Aug;32(8):570-9. doi: 10.1002/da.22384. Epub 2015 Jun 26. PMID 26115513
- See also: The trauma program of the anxiety disorders clinic of New York State Psychiatric Institute/Columbia University. Click here for more information about this study: — http://www.columbiatrauma.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Started | 18 | 18
Completed | 6 | 3
Not Completed | 12 | 15
Not completed — Adverse Event | 4 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.7) | 42.4 (13.3) | 40.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  white | 4 | 5 | 9
  black | 4 | 3 | 7
  other | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — Measures severity of depression on scale from 0 (not depressed) to 50 (most severe).
  units on a scale | 20.8 (6.2) | 20.4 (5.9) | 20.6 (6.0)
Posttraumatic Stress Disorder Checklist [Mean (Standard Deviation); unit: units on a scale] — Measures severity of posttraumatic stress disorder symptoms from 17 (mildest) to 85 (most severe).
  units on a scale | 58.9 (11.0) | 60.0 (10.5) | 59.5 (10.8)
Quality of Life Enjoyment and Satisfaction Scale [Mean (Standard Deviation); unit: units on a scale] — Measures quality of life from 16 (lowest quality) to 80 (greatest).
  units on a scale | 39.1 (13.6) | 41.4 (13.5) | 40.2 (13.4)
Medical Outcomes Study Short Form 12 - Physical [Mean (Standard Deviation); unit: units on a scale] — Measures level of physical functioning from 0 (worst) to 100 (best).
  units on a scale | 43.9 (9.8) | 41.4 (10.6) | 42.7 (10.1)
Medical Outcomes Study Short Form 12 - Mental [Mean (Standard Deviation); unit: units on a scale] — Measures level of mental functioning from 0 (worst) to 100 (best).
  units on a scale | 30.3 (13.5) | 30.4 (10.0) | 30.4 (11.7)
Pittsburgh Sleep Quality Index Global [Mean (Standard Deviation); unit: units on a scale] — Measures severity of sleep impairment from 0 (least impairment) to 21 (most severe).
  units on a scale | 11.5 (4.9) | 12.8 (3.1) | 12.1 (4.1)
Pittsburgh Sleep Quality Index Addendum for PTSD [Mean (Standard Deviation); unit: units on a scale] — Measure severity of sleep impairment related to posttraumatic stress disorder symptoms on a scale from 0 (least impairment) to 100 (most impairment)
  units on a scale | 10.0 (4.9) | 11.2 (5.6) | 10.6 (5.2)
Clinician Administered PTSD Scale [Mean (Standard Deviation); unit: units on a scale] — Measures severity of posttraumatic stress disorder symptoms from 0 (least severe) to 136 (most severe).
  units on a scale | 77.9 (19.5) | 81.3 (12.2) | 79.6 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Severity
Description: PTSD severity will be measured by the Clinician-Administered Posttraumatic Stress Disorder Scale, from 0 (least severe) to 136 (most severe).
Time Frame: up to 24 weeks
Population: intention to treat sample
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
units on a scale | 23.8 (17.4) | 34.6 (17.7)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis

2. Primary Outcome: Time to Discontinuation of Study Treatment
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
days | 95.2 (73.1) | 90.0 (14.8)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.82, t-test, 2 sided

3. Secondary Outcome: Alternative Measure of PTSD Severity
Description: as measured by the Short Posttraumatic Stress Disorder Rating Interview, which rates severity of PTSD from 0 (least severe) to 32 (most severe)
Time Frame: up to 24 weeks
Population: completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 9 | 6
units on a scale | 3.4 (2.9) | 6.7 (5.0)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = .14, t-test, 2 sided

4. Secondary Outcome: PTSD Self-rated Severity
Description: as measured by the PTSD Checklist which rates severity of PTSD from 17 (least severe) to 85 (most severe).
Time Frame: up to 24 weeks
Population: completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 9 | 9
units on a scale | 33.2 (18.4) | 39.2 (18.2)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = .50, t-test, 2 sided

5. Secondary Outcome: Depression Severity
Description: as measured by the 17-item Hamilton Rating Scale for Depression, which rates severity of depression on a scale from 0 (least depression) to 50 (greatest depression).
Time Frame: up to 24 weeks
Population: intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
units on a scale | 6.4 (6.1) | 11.6 (6.4)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis

6. Secondary Outcome: Response Status
Description: Responders defined by Clinician Administered Posttraumatic Stress Disorder Scale total score decreased by at least 30% compared with baseline and Clinical Global Impression improvement score of =1 or 2 at endpoint
Time Frame: up to 24 weeks
Population: intent to treat
Measure: Number; unit: percentage of subjects
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
percentage of subjects | 56 | 22
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.31, Mixed Models Analysis; Odds Ratio (OR) = 1.8

7. Secondary Outcome: Remission Status
Description: Remitter as defined by Clinician Administered Posttraumatic Stress Disorders Scale total score <20 at endpoint
Time Frame: up to 24 weeks
Population: intent to treat
Measure: Number; unit: percentage of subjects
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
percentage of subjects | 39 | 11
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis; Odds Ratio (OR) = 4.7, 95% CI 2-sided [1.1 to 19.9]

8. Secondary Outcome: Adverse Effects
Description: as assessed by Side Effect Checklist
Time Frame: up to 24 weeks
Population: intent to treat
Measure: Number; unit: percentage of subject dropped due to AEs
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
percentage of subject dropped due to AEs | 22.2 | 33.3
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.14, Chi-squared

9. Secondary Outcome: Sleep Quality
Description: as measured by Pittsburgh Sleep Quality Index, which rates severity of impairment in sleep quality from 0 (least impaired) to 21 (most impaired).
Time Frame: up to 24 weeks
Population: intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
units on a scale | 4.4 (4.2) | 9.1 (4.9)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis

10. Secondary Outcome: Sexual Functioning
Description: as measured by Arizona Sexual Experiences Scale, which rates impairment in sexual functioning from 5 (least impaired) to 30 (most impaired).
Time Frame: up to 24 weeks
Population: intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Number analyzed (Participants) | 18 | 18
units on a scale | 16.3 (4.3) | 17.4 (8.1)
Statistical Analysis 1: Comparison: Sertraline and Mirtazapine vs Sertraline and Sugar Pill; Test type: Superiority or Other; p = 0.65, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Sertraline and Mirtazapine | Sertraline and Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 18/18 | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sertraline and Mirtazapine (N=18) | Sertraline and Sugar Pill (N=18)
headache (Nervous system disorders) | 4 | 3
heartburn (Gastrointestinal disorders) | 5 | 3
nausea (Gastrointestinal disorders) | 2 | 8
emesis (Gastrointestinal disorders) | 2 | 3
decreased appetite (Gastrointestinal disorders) | 3 | 5
increased appetite (Gastrointestinal disorders) | 9 | 2
dry mouth (Gastrointestinal disorders) | 3 | 5
constipation (Gastrointestinal disorders) | 3 | 5
diarrhea (Gastrointestinal disorders) | 6 | 5
sweating (Skin and subcutaneous tissue disorders) | 4 | 5
skin problems (Skin and subcutaneous tissue disorders) | 4 | 1
bruising (Blood and lymphatic system disorders) | 0 | 1
restlessness (Nervous system disorders) | 2 | 1
tremor (Nervous system disorders) | 5 | 5
nervousness (Nervous system disorders) | 1 | 1
incoordination (Nervous system disorders) | 3 | 2
insomnia (Nervous system disorders) | 2 | 2
fatigue (General disorders) | 1 | 6
somnolence (Nervous system disorders) | 6 | 5
decreased libido (men) (Reproductive system and breast disorders) | 0/6 | 3/7
decreased libido (women) (Reproductive system and breast disorders) | 5/12 | 3/11
sexual dysfunction (men) (Reproductive system and breast disorders) | 0/6 | 3/7
sexual dysfunction (women) (Reproductive system and breast disorders) | 1/12 | 2/11
urinary dysfunction (Renal and urinary disorders) | 5 | 5
blurry vision (Eye disorders) | 4 | 2
lightheadedness (Nervous system disorders) | 9 | 4
forgetfulness (Nervous system disorders) | 4 | 4
impaired concentration (Nervous system disorders) | 2 | 4
apathy (Nervous system disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
small sample due to low recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No